CLINICAL TRIAL: NCT01956513
Title: Etude ADC Apport de l'IRM Dans l'évaluation du Coefficient de Diffusion Apparent et prédiction de la réponse à la chimiothérapie néoadjuvante Dans le Cancer du Sein
Brief Title: Contribution of MRI in the Evaluation of Apparent Diffusion Coefficient and Prediction of Response to Neoadjuvant Chemotherapy in Breast Cancer
Acronym: ADC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We have finally no financial support and any patients have been included.
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Etude ADC
Record Dates: First submitted 2012-03-16; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Assess the Variation of Apparent Diffusion Coefficient
Keywords: ADC; breast cancer; complete pathological response
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MRI (Magnetic resonance imaging) — MRI will be realised at the beginning of the study, after a cycle of chemotherapy or at changement of sequence and at the end of chemotherapy.

SUMMARY:
The main objective of the study is to assess the sensitivity and the specificity of the variation of apparent diffusion coefficient for prediction, after a course of neoadjuvant chemotherapy or after modification of the treatment sequence, the pathological response at the end of chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years.
* Patient suffering from a breast tumor, regardless of the stage and size
* Patient requiring neoadjuvant chemotherapy
* Patient has the ability to undergo 18F-FDG-PET at baseline, at end of cycle 1 and at the end of neoadjuvant treatment before surgery
* Compulsory affiliation to a social security system.
* Obtaining informed consent in writing, signed and dated.

Exclusion Criteria:

* Patient with cognitive or psychiatric disorders.
* Patient deprived of liberty by a court or administrative.
* Patient with signs against the achievement of MRI, mammography and ultrasound
* Patient metastatic
* Patient with prior chemotherapy, radiotherapy and hormone therapy for her breast cancer
* Pregnant women, current lactation
* Patient suffering from uncontrolled diabetes (> 11 mmol / L)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Variation of apparent diffusion coefficient before / after a cycle of neoadjuvant chemotherapy or before / after modification of the treatment sequence and correlated with histologic response | One year

CONTACTS AND LOCATIONS:
Overall Officials: Anne BAILLY, MD, Principal Investigator — Centre Jean Perrin